CLINICAL TRIAL: NCT02958267
Title: Investigation of Mesenchymal Stem Cell Therapy for the Treatment of Osteoarthritis of the Knee: Effect on Pain and Quality of Life
Brief Title: Investigation of Mesenchymal Stem Cell Therapy for the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, Joseph Ruane, Principal Investigator - Medical Director, McConnell Heart Health Center, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OH1-16-00672
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; regenerative medicine; orthobiologics; cellular therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- BMAC injection and PRP injection (Experimental): Injection of bone marrow aspirate concentrate (BMAC) withdrawn from a bone near the hip into the knee joint (intra-articular) immediately followed by an injection of platelet-rich plasma (PRP) into the knee joint.
  Interventions: Biological: BMAC injection; Biological: PRP injection
- Gel-One® hyaluronate injection (Active Comparator): Gel-One® is an hyaluronate gel used in the treatment of knee osteoarthritis by injection into the knee joint (intra-articular).
  Interventions: Device: Gel-One® hyaluronate injection

INTERVENTIONS:
Biological: BMAC injection — 60mL of bone marrow will be collected from a bone near the hip. Approximately 5-6mL of the bone marrow aspirate concentrate is then used for injection, under ultrasound guidance, into the target knee by the study physician.
  Arms: BMAC injection and PRP injection
Biological: PRP injection — 60mL of venous blood will be withdrawn from either arm. Approximately 4-5 ml of platelet-rich plasma will be introduced under ultrasound guidance to the subject's target knee by the study physician.
  Arms: BMAC injection and PRP injection
Device: Gel-One® hyaluronate injection — Patients will receive a single injection of Gel-One® (3 ml syringe of Gel-One® - 1% solution [10 mg/mL], 30mg total hyaluronan) into the target knee. Injections will be performed by the study physician under real-time dynamic ultrasound guidance.
  Arms: Gel-One® hyaluronate injection

SUMMARY:
The purpose of this study is to determine the clinical response to autologous bone marrow aspirate concentrate (BMAC) and platelet-rich plasma (PRP) injections for knee osteoarthritis with respect to pain, function, and quality of life at up to 1 year following the intervention. Specifically, the clinical response will be compared to baseline and a control group treated with a Gel-One® hyaluronate injection to the target knee.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 40 to 70 years old
2. Diagnosed with knee osteoarthritis based on the American College of Rheumatology criteria including symptomatic reports and radiographic findings
3. Kellgren-Lawrence grade 1-3 based on a radiograph within 6 months of presentation to the clinic
4. Symptomatic evidence of tibiofemoral osteoarthritis for ≥6 months
5. Average numeric pain rating of 4 - 8 on a scale of zero to 10 (defined as moderate level) over the past week
6. Previous trial of 6 weeks minimum of conservative therapy including physical therapy, weight loss, anti-inflammatory medication, or injection therapy

Exclusion Criteria:

1. Grade 4 knee osteoarthritis according to the Kellgren-Lawrence scale
2. History of intraarticular viscosupplementation or steroid injection in the target knee in the past 6 months at the time of the baseline visit or intraarticular injection planned during the trial
3. History of arthroscopic surgery in the target knee in the past 12 months at the time of presentation to the clinic or planned surgery during the trial period (e.g., scheduled for/awaiting arthroscopy or a knee replacement procedure)
4. Bilateral knee osteoarthritis (unless the contralateral knee involvement is limited to radiographic osteoarthritis and not symptomatic)
5. Ipsilateral (same side) or contralateral (opposite side) symptomatic osteoarthritis of hip or ankle
6. Clinically apparent tense effusion or other acute inflammation of the target knee at the time of presentation to the clinic
7. Active infection of either lower extremity such as cellulitis or any skin disease or infection in the area where BMAC is aspirated, blood is drawn, or an injection is given
8. History of diagnosis of any of the following: 1) septic osteoarthritis of any joint, 2) inflammatory arthropathy such as rheumatoid arthritis, gout, pseudogout, lupus, crystalline arthropathy, chondrocalcinosis and other rheumatology diagnoses
9. Cruciate/collateral knee ligament instability, ligament laxity, or meniscal instability of the target knee
10. Significant alignment deformity such as varus/valgus of the target knee in the judgment of the investigator
11. Currently pregnant, nursing, or planning to become pregnant during the trial period
12. Previous or known allergic reaction or hypersensitivity to heparin; sodium citrate; hyaluronan products or specifically Gel-One®; cinnamon; bird products such as feathers, eggs, or poultry; avian proteins
13. Not suitable for BMAC tissue allograft injection per physician (e.g., blood dyscrasia)
14. Unable to be prescribed stable dose of NSAIDs and/or tramadol based on medical history as ad lib use of over-the-counter analgesics will be allowed in both groups after treatment
15. Current cigarette smoker
16. Unable to give informed consent
17. Non-English speaking

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Ruane, DO, Principal Investigator — Medical Director, McConnell Heart Health Center
Locations (1):
- McConnell Spine, Sport, and Joint Physicians, Columbus, Ohio, United States

REFERENCES:
- [Derived] Ruane JJ, Ross A, Zigmont V, McClure D, Gascon G. A Single-Blinded Randomized Controlled Trial of Mesenchymal Stem Cell Therapy for the Treatment of Osteoarthritis of the Knee with Active Control. J Stem Cells Regen Med. 2021 Jan 2;17(1):3-17. doi: 10.46582/jsrm.1701002. eCollection 2021. PMID 34434003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of participants to be treated was capped at 30 participants. However, the approved protocol allowed enrollment of up to 45 participants to achieve a treatment group of 30 participants.
Pre-assignment Details: Based on the recruitment details stated, if a participant enrolled but subsequently withdrew or was withdrawn prior to treatment, another participant was enrolled in order to achieve a number of 30 participants who were treated within the study. Per protocol, consented patients could include up to 45 if needed to achieve 30 treated participants.
Period: Enrollment
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
Started | 17 | 15
Completed | 17 | 15
Not Completed | 0 | 0
Period: Enrollment to Actual Treatment Complete
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
Started | 17 | 15
Completed | 15 | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Follow-up Visits
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
Started | 15 | 15
3 Month Follow-up | 15 | 15
6 Month Follow-up | 14 | 14
12 Month Follow-up | 13 | 14
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — Additional treatment pursued | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.06 (9.14) | 58.60 (8.05) | 58.31 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 10 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.19 (5.19) | 29.21 (7.05) | 29.20 (6.03)
Previous surgery on target knee knee [Count of Participants; unit: Participants]
  No | 7 | 6 | 13
  Yes | 10 | 9 | 19
Previous injection on target knee [Count of Participants; unit: Participants]
  No | 6 | 8 | 14
  Yes | 11 | 7 | 18
Previous physical therapy on target knee [Count of Participants; unit: Participants]
  No | 4 | 9 | 13
  Yes | 13 | 6 | 19
Onset/course of target knee [Count of Participants; unit: Participants]
  Traumatic | 5 | 6 | 11
  Insidious | 12 | 9 | 21
Kellgren-Lawrence grade (n, %) [Count of Participants; unit: Participants] — PI assigned grade using criteria from source on p.42: Schiphof D, Boers M, Bierma-Zeinstra SMA. Differences in descriptions of kellgren and lawrence grades of knee osteoarthritis. Annals of the rheumatic diseases. 2008;67(7):1034-1034
  1. Doubtful narrowing of joint space and possible osteophytic lipping
  2. Definite osteophytes and possible narrowing of joint space
  3. Moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends
  4. Large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends
  Participants
    Grade 1 | 5 | 2 | 7
    Grade 2 | 6 | 8 | 14
    Grade 3 | 6 | 5 | 11
KOOS Pain [Mean (Standard Deviation); unit: units on a scale] — The Knee injury and Osteoarthritis Outcome Score consists of 5 subscales (i.e., pain, symptoms, function in activities of daily living, function in sport and recreation, and knee-related quality of life) developed to assess change over time in those with primary OA or knee injuries resulting in post-traumatic OA (Roos & Lohmander, 2003). A change in 10 points is considered clinically important (Roos & Lohmander, 2003). Scores are reported on a scale of 0-100 with 100 representing the best possible score.
  units on a scale | 60.82 (15.05) | 63.33 (17.72) | 62.00 (16.13)
KOOS Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Knee injury and Osteoarthritis Outcome Score consists of 5 subscales (i.e., pain, symptoms, function in activities of daily living, function in sport and recreation, and knee-related quality of life) developed to assess change over time in those with primary OA or knee injuries resulting in post-traumatic OA (Roos & Lohmander, 2003). A change in 10 points is considered clinically important (Roos & Lohmander, 2003). Scores are reported on a scale of 0-100 with 100 representing the best possible score.
  units on a scale | 66.54 (16.01) | 68.80 (15.69) | 67.59 (15.65)
KOOS ADLs [Mean (Standard Deviation); unit: units on a scale] — The Knee injury and Osteoarthritis Outcome Score consists of 5 subscales (i.e., pain, symptoms, function in activities of daily living, function in sport and recreation, and knee-related quality of life) developed to assess change over time in those with primary OA or knee injuries resulting in post-traumatic OA (Roos & Lohmander, 2003). A change in 10 points is considered clinically important (Roos & Lohmander, 2003). Scores are reported on a scale of 0-100 with 100 representing the best possible score.
  units on a scale | 68.59 (17.98) | 70.13 (18.34) | 69.31 (17.87)
KOOS Sport & Recreation [Mean (Standard Deviation); unit: units on a scale] — The Knee injury and Osteoarthritis Outcome Score consists of 5 subscales (i.e., pain, symptoms, function in activities of daily living, function in sport and recreation, and knee-related quality of life) developed to assess change over time in those with primary OA or knee injuries resulting in post-traumatic OA (Roos & Lohmander, 2003). A change in 10 points is considered clinically important (Roos & Lohmander, 2003). Scores are reported on a scale of 0-100 with 100 representing the best possible score.
  units on a scale | 31.47 (23.57) | 39.67 (21.59) | 35.31 (22.68)
KOOS Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The Knee injury and Osteoarthritis Outcome Score consists of 5 subscales (i.e., pain, symptoms, function in activities of daily living, function in sport and recreation, and knee-related quality of life) developed to assess change over time in those with primary OA or knee injuries resulting in post-traumatic OA (Roos & Lohmander, 2003). A change in 10 points is considered clinically important (Roos & Lohmander, 2003). Scores are reported on a scale of 0-100 with 100 representing the best possible score.
  units on a scale | 36.18 (18.50) | 38.47 (15.94) | 37.25 (17.11)
NPRS [Mean (Standard Deviation); unit: units on a scale] — The 11-point Numeric Pain Rating Scale (NPRS) is commonly used to assess the level and change of patient reported pain over time. Pain is rated from 0 to 10 with zero representing 'no pain' and 10 representing 'worst imaginable pain' (Farrer, Young, LaMoreaux, Werth, & Poole, 2001). A 2-point or 30-33% reduction has been established as a clinically important difference in populations with chronic musculoskeletal pain, including knee OA (Farrer, Young, LaMoreaux, Werth, & Poole, 2001; Salaffi, Stancati, Silvestri, Ciapetti, & Grassi, 2004).
  units on a scale | 4.59 (1.84) | 4.20 (1.70) | 4.41 (1.76)
PROMIS Global Health Physical Score [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System (PROMIS®) Global Health scale v1.1 contains 10 questions and produces two subscale scores: Global Physical Health (GPH) and Global Mental Health (GMH) (Hays, Bjorner, Revicki, Spritzer, & Cella, 2009). Each subscale produces a raw score that is converted to a T score such that an average patient in the United States would have a subscale T score of 50 with a standard deviation of 10 points ("Global Health: A Brief Guide to the PROMIS® Global Health Instruments", 2017).
  units on a scale | 44.62 (7.61) | 48.23 (7.99) | 46.31 (7.88)
PROMIS Global Health Mental Score [Mean (Standard Deviation); unit: units on a scale] — The Patient Reported Outcomes Measurement Information System (PROMIS®) Global Health scale v1.1 contains 10 questions and produces two subscale scores: Global Physical Health (GPH) and Global Mental Health (GMH) (Hays, Bjorner, Revicki, Spritzer, & Cella, 2009). Each subscale produces a raw score that is converted to a T score such that an average patient in the United States would have a subscale T score of 50 with a standard deviation of 10 points ("Global Health: A Brief Guide to the PROMIS® Global Health Instruments", 2017).
  units on a scale | 51.88 (5.02) | 51.90 (9.36) | 51.89 (7.25)

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score
Description: Subscales include pain, symptoms, function in activities of daily living, function in sport and recreation, and knee-related quality of life. Each subscale is 0-100 with 100 indicating the best possible score.
Time Frame: Change from baseline to 3, 6, and 12 months post-treatment
Population: One participant in the BMAC injection and PRP injection group withdrew prior to the 6 month follow-up and another prior to the 12 month follow-up both due to the pursuit of an additional treatment option. One participant in the hyaluronate injection group withdrew prior to the 6 month follow-up due to pursuit of an additional treatment option.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
Number analyzed (Participants) | 15 | 15
score on a scale
  KOOS Pain (3 months) | 16.71 [6.71 to 26.71] | 10.93 [5.15 to 16.71]
  KOOS Symptoms (3 months) | 14.00 [4.38 to 23.63] | 10.47 [3.48 to 17.45]
  KOOS ADL (3 months) | 15.35 [5.10 to 25.59] | 12.47 [5.97 to 18.96]
  KOOS Sport (3 months) | 29.46 [13.02 to 45.91] | 30.07 [18.71 to 41.43]
  KOOS QOL (3 months) | 21.02 [9.03 to 33.01] | 21.27 [11.10 to 31.43]
  KOOS Pain (6 months): number analyzed (Participants) | 14 | 14
  KOOS Pain (6 months) | 20.03 [10.71 to 29.36] | 12.52 [3.16 to 21.89]
  KOOS Symptoms (6 months): number analyzed (Participants) | 14 | 14
  KOOS Symptoms (6 months) | 14.26 [4.70 to 23.81] | 12.41 [5.45 to 19.37]
  KOOS ADLs (6 months): number analyzed (Participants) | 14 | 14
  KOOS ADLs (6 months) | 18.13 [9.00 to 27.25] | 14.94 [5.98 to 23.90]
  KOOS Sport (6 months): number analyzed (Participants) | 14 | 14
  KOOS Sport (6 months) | 34.89 [19.90 to 49.88] | 31.62 [16.41 to 46.82]
  KOOS QOL (6 months): number analyzed (Participants) | 14 | 14
  KOOS QOL (6 months) | 24.97 [14.51 to 35.42] | 24.18 [10.99 to 37.36]
  KOOS Pain (12 months): number analyzed (Participants) | 13 | 14
  KOOS Pain (12 months) | 23.48 [14.85 to 32.12] | 12.67 [2.62 to 22.71]
  KOOS Symptoms (12 months): number analyzed (Participants) | 13 | 14
  KOOS Symptoms (12 months) | 18.01 [10.29 to 25.72] | 8.20 [0.33 to 16.73]
  KOOS ADLs (12 months): number analyzed (Participants) | 13 | 14
  KOOS ADLs (12 months) | 19.10 [9.52 to 28.68] | 11.87 [2.05 to 21.68]
  KOOS Sport (12 months): number analyzed (Participants) | 13 | 14
  KOOS Sport (12 months) | 39.07 [22.00 to 56.13] | 26.05 [13.16 to 38.93]
  KOOS QOL (12 months): number analyzed (Participants) | 13 | 14
  KOOS QOL (12 months) | 27.44 [17.61 to 37.27] | 21.46 [8.33 to 34.60]

2. Secondary Outcome: Numeric Pain Rating Scale
Description: Scale from 0-10 with 0 representing "no pain" and 10 representing "worst imaginable pain"
Time Frame: Change from baseline to 3, 6, and 12 months post-treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
Number analyzed (Participants) | 15 | 15
score on a scale
  NPRS (3 months) | -1.92 [-3.27 to -0.57] | -1.87 [-2.76 to -0.97]
  NPRS (6 months): number analyzed (Participants) | 14 | 14
  NPRS (6 months) | -2.45 [-3.60 to -1.28] | -1.77 [-2.55 to -0.99]
  NPRS (12 months): number analyzed (Participants) | 13 | 14
  NPRS (12 months) | -3.13 [-3.96 to -2.29] | -1.56 [-2.59 to -0.53]

3. Secondary Outcome: Patient Reported Outcome Measurement Information System Global Health Scores
Description: The Patient Reported Outcomes Measurement Information System (PROMIS®) Global Health scale v1.1 contains 10 questions and produces two subscale scores: Global Physical Health (GPH) and Global Mental Health (GMH) (Hays, Bjorner, Revicki, Spritzer, & Cella, 2009). Each subscale produces a raw score that is converted to a T score such that an average patient in the United States would have a subscale T score of 50 with a standard deviation of 10 points ("Global Health: A Brief Guide to the PROMIS® Global Health Instruments", 2017). A score higher than the mean indicates a more desirable score, and vice versa. A positive change score indicates an improvement, while a negative change score indicates a decline in score value.
Time Frame: Change from baseline to 3, 6, and 12 months post-treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
Number analyzed (Participants) | 15 | 15
score on a scale
  PROMIS Physical Health (3 months) | 4.62 [0.84 to 8.41] | 0.59 [-3.76 to 4.94]
  PROMIS Mental Health (3 months) | -2.18 [-3.87 to -0.48] | -0.65 [-5.13 to 5.83]
  PROMIS Physical Health (6 months): number analyzed (Participants) | 14 | 14
  PROMIS Physical Health (6 months) | 6.76 [3.63 to 9.89] | 3.50 [0.16 to 6.83]
  PROMIS Mental Health (6 months): number analyzed (Participants) | 14 | 14
  PROMIS Mental Health (6 months) | -0.01 [-3.25 to 3.23] | 2.24 [-0.54 to 5.03]
  PROMIS Physical Health (12 months): number analyzed (Participants) | 13 | 14
  PROMIS Physical Health (12 months) | 4.77 [1.99 to 7.54] | 3.26 [-0.36 to 6.88]
  PROMIS Mental Health (12 months): number analyzed (Participants) | 13 | 14
  PROMIS Mental Health (12 months) | 0.07 [-2.64 to 2.77] | 3.01 [-0.40 to 6.42]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent/enrollment through approximately 12 months following each participant's treatment date or until participant withdrawal, whichever occurred first.
Description: Included in this report are any adverse events considered unexpected and therefore not listed on the research protocol and informed consent documents as common or likely, less common, or rare risks.
Arm/Group | BMAC Injection and PRP Injection | Gel-One® Hyaluronate Injection
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 1/17 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMAC Injection and PRP Injection (N=17) | Gel-One® Hyaluronate Injection (N=15)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT02958267/Prot_SAP_000.pdf